CLINICAL TRIAL: NCT00191542
Title: A Randomised, Double Blind Placebo Controlled Study of the Broader Efficacy of Atomoxetine Hydrochloride in the Treatment of Attention-Deficit/Hyperactivity Disorder (ADHD) in Swedish Children and Adolescents
Brief Title: Atomoxetine vs Placebo in the Treatment of ADHD in Swedish Children and Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6671; B4Z-SO-LY15
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2006-10-11 (Estimated); Status verified 2006-10

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

INTERVENTIONS:
Drug: Atomoxetine
Drug: Placebo

SUMMARY:
Comparison of the effect of Atomoxetine and psychoeducation with placebo and psychoeducation after 10 weeks of treatment

ELIGIBILITY:
Inclusion Criteria:

* Meet the criteria for ADHD of the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) as well as severity criteria. Diagnosis is assessed by the investigator's clinical evaluation as well as administration of the K-SADS-PL structured interview.
* Meet a symptom severity threshold of 1.5 standard deviations above age and sex norms for their diagnostic subtype on the ADHDRS-IV-Parent: Investigator-Administered and Scored (ADHDRS-IV-Parent:Inv) This severity threshold must be met at Visit 1 and maintained at Visit 2.
* Be at least 7 years of age, but not yet have reached their 16th birthday prior to Visit 1, when informed consent is obtained.
* For female subjects of child-bearing potential only, test negative for pregnancy at the time of enrollment based on a urine pregnancy test and agree to use a reliable method of birth control.

Exclusion Criteria:

* Weigh less than 20 kg at study entry
* Have a documented history of Bipolar Disorder or any history of psychosis or pervasive development disorder (autistic spectrum disorder).
* Are pregnant or breastfeeding.
* Are at serious suicidal risk as assessed by the investigator.
* Have been treated previously for ADHD with pyschostimulants such as Methylphenidate or Ritalin

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100
Dates: Start 2005-03; Study Completion 2006-08

PRIMARY OUTCOMES:
To test the hypothesis that atomoxetine and psychoeducation given for 10 weeks is superior to placebo and psychoeducation in improving overall
functioning of patients with ADHD as measured by the mean change in the total score of the Child Health and Illness Profile-Child Edition-Parent form (CHIP-CE-Parent form) domain Achievement.

SECONDARY OUTCOMES:
To compare the effects of atomoxetine and psychoeducation with those of placebo and psychoeducation at 10 weeks in patients with ADHD as measured by change in the CHIP-CE-Parent form domains Satisfaction, Comfort, Resilience, and Risk avoidance.
To compare the effects of atomoxetine and psychoeducation with those of placebo and psychoeducation at 10 weeks in patients with ADHD with regard to core ADHD symptoms, as measured by the ADHDRS total score.
To compare the effects of atomoxetine and psychoeducation with those of placebo and psychoeducation at 10 weeks in patients with ADHD with regard to severity of illness and improvement, as measured by the CGI-ADHD-S and CGI-ADHD-I.
To compare the effects of atomoxetine and psychoeducation with those of placebo and psychoeducation at 10 weeks in patients with ADHD with regard to self-perception, as measured by the "I Think I Am" ("Jag tycker jag ar") tool.
To compare the effects of atomoxetine and psychoeducation with those of placebo and psychoeducation at 10 weeks in patients with ADHD as measured by change in all twelve CHIP-CE-Parent form subdomains.
To compare the effects of atomoxetine and psychoeducation with those of placebo and psychoeducation at 10 weeks in patients with ADHD as measured by change in total CHIP-CE-Parent form score.
To compare the effects of atomoxetine and psychoeducation with those of placebo and psychoeducation at 10 weeks in patients with ADHD with regard to family stress, as measured by the Appraisals of Stress in Child-Rearing (ASCR).
To compare the effects of atomoxetine and psychoeducation with those of placebo and psychoeducation at 10 weeks in patients with ADHD with regard to family burden of illness, as measured by the FBIM.
To investigate the concurrent validity of the FBIM and the ASCR in order to test the validity of the former instrument in a Swedish population.
To assess whether the changes in scores on the aforementioned rating scales are maintained over the longer term (at week 17, 25, 37, and 49, respectively; for "I think I am" at week 49 only).
To investigate if the results are modified by comorbid and/or developmental problems as measured by the "Five to Fifteen" (FTF) and K-SADS.
To assess the long-term safety of atomoxetine.
To assess the utilization of resources and costs to families and society between atomoxetine and placebo
during the 10 week double blind treatment period and for each patient during the following open label extension period, using the Resource Utilization Questionnaire (RUQ)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (9):
- Sweden (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Gothenburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Huddinge
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Linköping
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Lund
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Mölnlycke
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Örebro
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Umeå
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Uppsala
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Vaxjo

REFERENCES:
- [Derived] Bangs ME, Wietecha LA, Wang S, Buchanan AS, Kelsey DK. Meta-analysis of suicide-related behavior or ideation in child, adolescent, and adult patients treated with atomoxetine. J Child Adolesc Psychopharmacol. 2014 Oct;24(8):426-34. doi: 10.1089/cap.2014.0005. Epub 2014 Jul 14. PMID 25019647